CLINICAL TRIAL: NCT03942289
Title: Investigating the Noradrenergic System in the Living Human Brain With Hybrid Molecular Functional Imaging
Brief Title: Human Aging and in Vivo Noradrenergic System
Acronym: NA_PET_MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL18_0409; 2018-003999-13 (EudraCT Number)
Record Dates: First submitted 2019-04-11; First posted 2019-05-08 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Parkinson Disease
Keywords: Human; Aging; Behavior; Noradrenergic system; Positron Emission Tomography; Magnetic Resonance Imaging
MeSH Terms: conditions — Parkinson Disease; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy controls (Experimental)
  Interventions: Other: The role of the noradrenergic system across the life span (Healthy Subjects)
- Parkinson disease (Experimental)
  Interventions: Other: The role of the noradrenergic system across the life span (Parkinson's Disease Subjects)

INTERVENTIONS:
Other: The role of the noradrenergic system across the life span (Healthy Subjects) — A sample (n=90) of balanced distribution of healthy males and females within a continuous segment of the adult life span from 20 to 80 years old will be recruited, with approximately 7 males and 7 females subjects for each decade of age. Each participant will undergo 1) a neuropsychological examination, 2) an olfactory screening and 3) a 90 min 11C-Yohimbine positron emission tomography (PET)/magnetic resonance imaging (MRI) scan in a resting state.
  Arms: Healthy controls
Other: The role of the noradrenergic system across the life span (Parkinson's Disease Subjects) — Three groups of Parkinson Disease (PD) patients (each of them n=15) will be studied according to the duration and stage of the disease: early stage (the same group in Task 2); mid stage (5-7 years of disease duration; Hoehn and Yahr in Off 2-3); late stage (7-10 years of disease duration; Hoehn and Yahr in Off 3-4).
  Arms: Parkinson disease

SUMMARY:
The main goal of this research proposal is to provide, for the first time in humans, a wider understanding of the role of the noradrenergic system both in health and illness (Parkinson's disease) through the use of a newly developed radiotracer (11Carbon [11C]Yohimbine) visualizing alpha-2 (α2) adrenergic receptors (AR) combined with cutting-edge technology, the hybrid positron emission tomography (PET)/magnetic resonance imaging (MRI) scanner. The secondary aim of this study will be to determine whether the expected age- and Parkinson's disease (PD)-related changes in the noradrenergic system are paralleled by changes in neuropsychological performances (such as cognitive, motor and/or olfactory abilities).

ELIGIBILITY:
Inclusion Criteria for the healthy controls:

* Age between 20 years and 80 years
* Weight between 40 kilograms (kg) and 95kg
* Without neurologic or psychiatric history
* Without head trauma history including loss of consciousness superior to 30 minutes.
* Affiliated to a social security or similar scheme
* Not subject to any legal protection measures
* Participant must have signed an informed consent document indicating that they understand the purpose of, and procedures required for, the study and are willing to participate in the study and comply with the study procedures and restrictions

Inclusion Criteria for the patients with Parkinson's disease:

* Age between 40 and 80 years old
* Weight between 40 kilograms (kg) and 95kg
* With an idiopathic Parkinson's disease (Dopa-sensitive)
* Without head trauma history including loss of consciousness superior to 30 minutes.
* Affiliated to a social security or similar scheme
* Not subject to any legal protection measures
* Participant must have signed an informed consent document indicating that they understand the purpose of, and procedures required for, the study and are willing to participate in the study and comply with the study procedures and restrictions

Exclusion Criteria:

* Subject with alcohol or substance abuse history
* Subject with somatic drug therapies
* Magnetic Resonance Imaging (MRI) contraindications (implanted or embedded metal objects in the head or body)
* Positron Emission Tomography (PET) contraindications
* Exposed to 1 millisievert or more of ionizing radiation in the year before the start of this study
* Subject unable to sign written consent for participation in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-06-29 (Estimated); Study Completion 2021-06-29 (Estimated)

PRIMARY OUTCOMES:
Positron Emission Tomography (PET) and Magnetic Resonance Imaging (MRI) measures | Day 1 -180 minutes
  Derived from the Positron Emission Tomography (PET) data, the binding potentials will be calculated using compartmental modelling techniques. Derived from the Magnetic Resonance Imaging (MRI) data.

SECONDARY OUTCOMES:
Global Cognitive Assessment | Day 2 - 10 minutes
  Measured with Montreal Cognitive Assessment. Outcome measure is between 0 and 30. A score of 26 or over is considered to be normal.
Memory Assessment | Day 2 - 20 minutes
  Measured with the 16-item Free and Cued Recall test. Outcome measure is the total immediate recall which is the sum of free and cued recall.
Working Memory Assessment | Day 2 - 20 minutes
  Measured with the Digit Span Memory test. Outcome measure is the total number of items correctly repeated.
Executive Functioning | Day 2 - 20 minutes
  Measured with the Trail Making test. Unit of measure is first seconds to perform the test, which will be converted in a percentile score and then number of errors made during the test.
Planning Functioning | Day 2 - 20 minutes
  Measured with the Tower of London test. Outcome measure is the total correct and total moves score.
Visuo-spatial Assessment | Day 2 - 20 minutes
  Measured by the Visual Object and Space Perception Battery. The study will use a selection of theses tests : incomplete letters (outcome measure is between 0 and 20; cut-off score = 16) and position discrimination (outcome measure is between 0 and 10; cut-off score = 7)
Depression Evaluation | Day 2 - 10 minutes
  Measured by the Beck Depression Inventory-II Questionnaire. Outcome measure is between 0 and 20 with a cut-off score = 13. A score higher than 14 indicates the presence of depression.
Anxiety Evaluation | Day 2 - 10 minutes
  Measured by the State-Trait Anxiety Inventory (STAI) form Y questionnaire. Outcome measure is between 20 and 80, with higher scores correlating with greater anxiety.
Praxic Abilities | Day 2 - 10 minutes
  Measured by the Mahieux Praxic test. Outcome measure is between 0 and 23.
Day time sleepiness evaluation | Day 2 - 5 minutes
  Measured by the Epworth Sleepiness Scale Questionnaire. Outcome measure is between 0 and 24 with a score between 0-8 indicating normal Daytime sleepiness, a score between 9-14 indicating mild sleep deficiency and a score above 15 an excessive daytime sleepiness.
Sleep Quality | Day 2 - 5 minutes
  Measured by the Pittsburgh Sleep Quality Index (PSQI). Outcome measure is between 0 and 21 with 0 indicating no sleep problem and 21 major sleep disorder.
Olfactory assessment : odor detection | Day 2 - 30 minutes
  The odor detection capability will be evaluated using a phenyl-ethyl alcohol (PEA) test. In this experiment, the detection threshold is obtained using a "staircase" procedure. Outcome measure is between 0 and 16 with higher score indicating better performance.
Olfactory assessment: odor discrimination | Day 2 - 30 minutes
  Odor discrimination capacity will be assessed by asking the participant to smell three bottles (two bottles contain the same odor, and the third contains a different smell). The test includes 16 triplets of odorous substances. Outcome measure is between 0 and 16 with higher score indicating better performance.
Olfactory assessment : odor identification | Day 2 - 30 minutes
  The odor identification capacity will be estimated by the European test of olfactory capacities (ETOC), a test based on 16 identifications. Outcome measure is between 0 and 16 with higher score indicating better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Chloé Laurencin, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Neurologique Pierre Wertheimer, Groupement Hospitalier Est, Bron, France